CLINICAL TRIAL: NCT06425796
Title: Impact of Maternal Adiposity on Maternal Iron Status and Requirements: a Randomised Intervention Study
Brief Title: Adiposity and Iron Requirements in Pregnancy
Acronym: ADIPREG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Solvotrin Therapeutics - Active Iron (Unknown); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FCBMS-23-259
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-03

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: Iron status; Iron Supplements; Pregnancy; Anaemia; Maternal obesity; Maternal Overweight; Body composition; Ferritin; Inflammation; Mental Health; Neonatal anaemia
MeSH Terms: conditions — Anemia; Pregnancy in Obesity; Inflammation; Psychological Well-Being; Anemia, Neonatal | interventions — Adiposity; Pregnancy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind: two or more parties are unaware of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron 25 (Active Comparator): Iron 25 (total 25 mg/d of iron): 2 supplements of 12.5 mg of elemental iron + 1 multivitamin supplement;
  Interventions: Dietary Supplement: Adiposity and Iron Requirements in Pregnancy (ADIPREG)
- IRON 50 (Active Comparator): Iron 50 (total 50 mg/d of iron): 2 supplements of 25 mg of elemental iron + 1 multivitamin supplement).
  Interventions: Dietary Supplement: Adiposity and Iron Requirements in Pregnancy (ADIPREG)

INTERVENTIONS:
Dietary Supplement: Adiposity and Iron Requirements in Pregnancy (ADIPREG) — Iron 25 arm will receive: two iron supplements containing 12.5 mg of elemental iron + 1 multivitamin supplement (they will receive a total of 3 supplements per day).
  Iron 50 arm will receive: two 25 mg elemental iron supplements + 1 multivitamin supplement (they will receive a total of 3 supplements per day).
  The multivitamin supplement will contain folic acid, vitamin B1, vitamin B2, vitamin B3, vitamin B5, vitamin B6, vitamin B12, vitamin C and vitamin D. In summary, each participant will receive 3 supplements per day and instructed to take the 3 supplements together, in the morning, with breakfast. Supplements will be given to the participants when they attend for their clinic appointment. The intervention will begin at 12 gestational weeks and continue until the baby is delivered.

SUMMARY:
This study aims to explore how body fat influences the response to either 25 or 50 mg of daily iron supplements during pregnancy. We will conduct a double-blind randomized controlled intervention study involving 312 pregnant women recruited from antenatal clinics in the Northern Trust Area. Participants will be randomly assigned to receive either 25 or 50 mg of iron per day from 12 weeks of pregnancy until delivery, using the Active Iron supplement brand. Blood samples will be collected at 12, 28 and 36 weeks gestation and umbilical cord blood will be collected at delivery. Anthropometric measurements will be taken at each visit, and participants will complete questionnaires on various aspects of health and lifestyle, mental health, gastrointestinal symptoms, and compliance.

DETAILED DESCRIPTION:
The main aim of this study is to investigate the influence of adiposity on the difference in response to 25 or 50 mg of daily iron supplementation during pregnancy. The primary aim is to determine the influence of maternal adiposity on adjusted maternal ferritin concentrations in response to 25 mg or 50 mg iron supplementation in pregnancy. The secondary outcomes of this study include: investigating the impact of maternal body fat on various maternal iron biomarkers (such as haemoglobin, soluble transferrin receptor, hepcidin, transferrin saturation, and other haematological markers) in response to either 25 mg or 50 mg iron supplementation during pregnancy, evaluating changes in adjusted ferritin concentrations and other iron markers throughout pregnancy relative to the dosage of iron supplementation received, determining the effect of maternal body fat on neonatal iron biomarkers in response to maternal iron supplementation, assessing changes in markers of inflammation in response to iron supplementation during pregnancy, and examine changes in mental health scores in response to iron supplementation during pregnancy.

This is a double-blind randomised controlled intervention study, in which 312 pregnant women with singleton pregnancy, without current complications, aged ≥ 18 years and BMI ≥ 18.5 kg/m2 will be recruited. Participants who are taking multivitamins will be included. They will be asked to discontinue any current supplementation. Pregnant women with anaemia, iron deficiency, high risk of iron overload, history of bariatric surgery, who are planning home birth, are currently involved in another research study, and those who cannot speak or understand English language will be excluded.

Blood samples and anthropometric and body composition measurements will be taken at different points in the pregnancy (12, 28, 36 gestational weeks) and an umbilical cord blood sample at the time of birth. Blood concentrations of iron and inflammation markers will be analysed. General, dietary intake and lifestyle information will be collected, through a Health and Lifestyle questionnaire and a 4-day diary. Additionally, participants will complete a questionnaire about their mental health and gastrointestinal symptoms. The compliance of the supplementation will be evaluated at each timepoint. Additionally, participants will receive a telephone call to evaluate possible adverse effects and compliance of the supplementation between the timepoints (18, 24 and 32 weeks of gestation). In the event that a participant has been prescribed iron treatment, anaemia diagnosis at any time during pregnancy or the occurrence of any adverse outcome such as miscarriage, the participant will be withdrawn from the study. Electronic forms prepared in RedCap will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:- Pregnant women

* Age ≥ 18 years
* BMI ≥18.5 kg/m2
* Without current pregnancy complications (for example, severe bleeding, Diabetes Mellitus, hyperemesis gravidarum, ectopic and molar pregnancies)
* At least 12 Gestational Week
* Singleton pregnancy confirmed with the first ultrasound scan
* Participants who are currently taking multivitamins will be included. They will be asked to discontinue any current supplementation.

Exclusion Criteria:

* Hb <110 g/L
* SF <30 μg/L
* High risk of iron overload (Hb >150 g/L, transferrin saturation >45% or SF> 150 μg/L)
* Participants with history of haematological, renal, liver, autoimmune disorders, malabsorptive syndromes
* Participants with history of bariatric surgery
* Participants who take steroids or anti-inflammatory treatments or drugs that affect gut absorption (proton-pump inhibitors)
* Planned home births
* Participants currently involved in another research study
* Multiple pregnancy
* Participants who do not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only female participants are being studied
Enrollment: 312 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
* - Adjusted maternal ferritin concentrations in response to iron supplementation (ng/mL) | 16, 24 and 28 weeks after baseline
  Assessed via electrochemiluminescence immunoassay "ECLIA".

SECONDARY OUTCOMES:
Hemoglobin (g/L) | 16, 24 and 28 weeks after baseline
  Assessed via Direct Current sheat flow method (Sysmex)
Red blood cell count (RBC) (10^12/L) | 16, 24 and 28 weeks after baseline.
  Assessed via Direct Current sheat flow method (Sysmex)
Mean cell haemoglobin (MCH) (pg | 16, 24 and 28 weeks after baseline.
  Assessed via Direct Current sheat flow method (Sysmex)
Mean cell volume (MCV) (fl) | 16, 24 and 28 weeks after baseline.
  Assessed via Direct Current sheat flow method (Sysmex)
Mean cell haemoglobin concentrations (MCHC) (g/dL) | 16, 24 and 28 weeks after baseline.
  Assessed via Direct Current sheat flow method (Sysmex)
Red cell distribution width (RDW) (%) | 16, 24 and 28 weeks after baseline.
  Assessed via Direct Current sheat flow method (Sysmex)
Transferrin (g/L) | 16, 24 and 28 weeks after baseline.
  Assessed via immunoturbidimety assay
Serum iron (umol/L) | 16, 24 and 28 weeks after baseline.
  Assessed via colorimetic assay
sTfR (ug/mL) | 16, 24 and 28 weeks after baseline.
  Assessed via ELISA
Hepcidin (pg/mL) | 16, 24 and 28 weeks after baseline.
  Assessed via ELISA
C-reactive protein (mg/mL) | 16, 24 and 28 weeks after baseline.
  Assessed via ELISA
Pro- anti- inflammatory biomarkers: IL-1 β, IL-6, IL-10, IL-22, IL-17, TNF- α, IFN- γ (fg/mL) | 16, 24 and 28 weeks after baseline.
  Assessed via sandwich immunoassay
Genetic variants of interest in relation to obesity and iron metabolism in response to iron supplementation. | 16, 24 and 28 weeks after baseline.
  Assessed via methylation analyses
Mental health score in response to iron supplementation | 16, 24 and 28 weeks after baseline
  CORE 10 questionnaire will be completed by each participant at each timepoint: CORE stands for "Clinical Outcomes in Routine Evaluation." The CORE-10 is a 10-item assesses psychological distress over the past week. The resulting score can be divided into categories with increasing severity: Healthy (0-5), low (6-10), mild (11-14), moderate (15-19), moderate-to-severe (20-24), and severe (25 and above). The score of this questionnaire will be collected as a numeric variable.

OTHER OUTCOMES:
Adjusted maternal ferritin concentrations in response to iron supplementation (ng/mL) | 16, 24 and 28 weeks after baseline
  Assessed via ELISA analyses for ferritin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Mary McCann, PhD, Study Director — University of Ulster
Locations (3):
- United Kingdom (3):
  - Causeway Hospital, Coleraine, Co Londonderry
  - Causeway Hospital, Coleraine, Co. Londonderry
  - Ulster University,Human Intervention Studies Unit,, Coleraine, Co. Londonderry

IPD SHARING:
Plan to Share IPD: No